CLINICAL TRIAL: NCT04209218
Title: Impact of Intraoperative Blood Pressure Management and Dexamethasone on Patient's Outcomes After Lung Cancer Surgery: A 2 × 2 Factorial Randomized Controlled Trial
Brief Title: Intraoperative Blood Pressure Management and Dexamethasone in Lung Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-234
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Surgery; Blood Pressure Management; Dexamethasone; Overall Survival; Postoperative Complications
Keywords: Lung Cancer; Radical Resection; Blood Pressure Management; Dexamethasone; Overall Survival; Postoperative Complications
MeSH Terms: conditions — Lung Neoplasms; Postoperative Complications | interventions — Dexamethasone; Glucocorticoids; Saline Solution

STUDY DESIGN:
Intervention Model Description: A 2 × 2 factorial randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: For dexamethasone administration, all participants, care providers, investigators, and outcomes assessors are masked. For blood pressure management, participants and outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Routine blood pressure management + placebo (Placebo Comparator): Blood pressure is maintained according to routine practice. Placebo (normal saline 2 ml) is administered before anesthesia induction.
  Interventions: Drug: Placebo; Other: Routine blood presure management
- Routine blood pressure management + dexamethasone (Experimental): Blood pressure is maintained according to routine practice. Dexamethasone (10 mg/2 ml) ia administered before anesthesia induction.
  Interventions: Drug: Dexamethasone; Other: Routine blood presure management
- Targeted blood pressure management + placebo (Experimental): Blood pressure is maintained within ±10% from baseline. Placebo (normal saline 2 ml) is administered before anesthesia induction.
  Interventions: Other: Targeted blood pressure management; Drug: Placebo
- Targeted blood pressure management + dexamethasone (Experimental): Blood pressure is maintained within ±10% from baseline. Dexamethasone (10 mg/2 ml) is administered before anesthesia induction.
  Interventions: Drug: Dexamethasone; Other: Targeted blood pressure management

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone (10 mg/2 ml) is administered before anesthesia induction.
  Other Names: Glucocorticoids
  Arms: Routine blood pressure management + dexamethasone; Targeted blood pressure management + dexamethasone
Other: Targeted blood pressure management — Blood pressure is maintained within ±10% from baseline.
  Arms: Targeted blood pressure management + dexamethasone; Targeted blood pressure management + placebo
Drug: Placebo — Placebo (2 ml normal saline) is administered before anesthesia induction.
  Other Names: Normal saline
  Arms: Routine blood pressure management + placebo; Targeted blood pressure management + placebo
Other: Routine blood presure management — Blood pressure is maintained according to routine practice.
  Arms: Routine blood pressure management + dexamethasone; Routine blood pressure management + placebo

SUMMARY:
Surgery is the front-line therapy for non-small cell lung cancer (NSCLC) but postoperative complications remains high and patients' long-term outcome is still challenging. In addition to surgery, anesthetic management particularly intraoperative blood pressure management and use of dexamethasone may affect patients' early and long-term outcomes after surgery for NSCLC. This study aims to investigate the impact of intraoperative blood pressure management and dexamethasone administration on early and long-term outcomes in patients undergoing surgery for lung cancer.

DETAILED DESCRIPTION:
Surgical resection is the main treatment for patients with non-small cell lung cancer (NSCLC) and continuous efforts have been made to evolve surgical strategies and techniques. It has been now been realized that perioperative period is characterized with profound changes and anesthesia management may also affect outcomes of patients after cancer surgery.

Even under well controlled conditions, blood pressure fluctuation frequently occurs during anesthesia and surgery. In previous studies, intraoperative hypotension was associated with increased risk of organ injuries (such as delirium, acute kidney injury, myocardial injury, and stroke) and higher 1-year mortality. Unpublished data showed that intraoperative hypotension was also associated with shortened long-term survival in patients after lung cancer surgery. In a recent trial, individualized intraoperative blood pressure management which avoided intraoperative hypotension decreased the incidence of postoperative organ injury when compared with routine practice. Avoiding intraoperative hypotension may also prolong survival after lung cancer surgery. However, evidences are lacking regarding this topic.

Dexamethasone is frequently used for prevention of postoperative nausea and vomiting. Studies showed that a single low-dose dexamethasone has anti-inflammatory effect and can regulate immune function. It has been shown that perioperative dexamethasone can improve analgesia after surgery. In retrospective studies, perioperative low-dose dexamethasone was associated with less wound infection and improved long-term survival in patients after surgeries for pancreatic and lung cancer. It is hypothesized that intraoperative dexamethasone may reduce postoperative complications and improve long-term survival after lung cancer surgery. Interventional studies are required to confirm this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Aged >50 years but <90 years.
* Diagnosed as resectable primary non-small cell lung cancer (stage IA-IIIA) and scheduled for radical surgery with an expected duration of >2 hours.
* Agree to participate in this study and sign the informed consent.

Exclusion Criteria:

* Clinical examinations suggest non-resectable lung cancer or patients scheduled for a biopsy surgery.
* Recurrent or metastatic lung cancer.
* History of cancer or complicated with cancer in other organs.
* Long-term exposure to glucocorticoids or other immunosuppressant(s) due to autoimmune disease or organ transplantation.
* Uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg); or requirement of vasopressors to maintain blood pressure.
* Persistent atrial fibrillation, or acute cardiovascular events (acute coronary syndrome, stroke, or congestive heart failure) within 3 months.
* Severe hepatic dysfunction (Child-Pugh C) or renal failure (requirement of renal replacement therapy).
* Any other circumstances considered unsuitable for study participation by attending physicians or investigators.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1988 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival after surgery | Up to 5 years after surgery
  Overall survival after surgery
Incidence of organ injury and complications within 5 days after surgery (sub-study). | Up to 5 days after surgery.
  Organ injury includes delirium, acute kidney injury and myocardial injury. Postoperative complications are generally defined as newly occurred medical conditions that are harmful to patients' recovery and required therapeutic intervention, i.e., grade II or above on the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Recurrence-free survival after surgery | Up to 5 years after surgery
  Recurrence-free survival after surgery
Cancer-specific survival after surgery | Up to 5 years after surgery
  Cancer-specific survival after surgery
Event-free survival after surgery | Up to 5 years after surgery
  Event-free survival after surgery
Rate of intensive care unit (ICU) admission after surgery (sub-study) | During the day of surgery
  Rate of ICU admission after surgery
Rate of ICU admission with endotracheal intubation after surgery (sub-study) | During the day of surgery
  Rate of ICU admission with endotracheal intubation after surgery
Duration of mechanical ventilation in ICU after surgery (sub-study) | Up to 30 days after surgery
  Duration of mechanical ventilation in ICU after surgery
Length of stay in ICU after surgery (sub-study) | Up to 30 days after surgery
  Length of stay in ICU after surgery
Incidence of organ injury within 5 days after surgery (sub-study) | Up to 5 days after surgery
  Organ injury includes delirium, acute kidney injury and myocardial injury. Delirium is assessed with the 3-minute diagnostic assessment for CAM-defined delirium (3D-CAM). Acute kidney injury is diagnosed according to the KDIGO (Kidney Disease: Improving Global Outcomes) criteria. Myocardial injury is diagnosed according to the serum cardiac troponin I level (higher than upper normal limit of the hospital's clinical laboratory).
Incidence of complications within 30 days after surgery (sub-study) | Up to 30 days after surgery
  Postoperative complications are defined as new-onset medical events that are harmful to patients' recovery and required therapeutic intervention, i.e., grade II or above on the Clavien-Dindo classification.
Length of stay in hospital after surgery (sub-study) | Up to 30 days after surgery
  Length of stay in hospital after surgery
Rate of 30-day all-cause mortality (sub-study) | Up to 30 days after surgery
  Death due to any cause within 30 days after surgery

OTHER OUTCOMES:
Overall survival after surgery in cancer patients | Up to 5 years after surgery
  Overall survival after surgery in cancer patients
Recurrence-free survival after surgery in cancer patients | Up to 5 years after surgery
  Recurrence-free survival after surgery in cancer patients
Cancer-specific survival after surgery in cancer patients | Up to 5 years after surgery
  Cancer-specific survival after surgery in cancer patients
Event-free survival after surgery in cancer patients | Up to 5 years after surgery
  Event-free survival after surgery in cancer patients
30-item quality of life in 1-, 2-, and 3-year survivors | At the end of the 1st, 2nd, and 3rd year after surgery
  Quality of life is assessed with the 30-item Core Quality of Life Questionnaire (QLQ-C30), which assess functioning and symptom scales. The score of each scale ranges from 0 to 100, with higher score indicating better function or worse symptom.
13-item quality of life in 1-, 2-, and 3-year survivors | At the end of the 1st, 2nd, and 3rd year after surgery
  Quality of life is assessed with the 13-item Quality of Life Questionnaire-Lung Cancer Module (QLQ LC-13), which assess symptom scales. The score of each scale ranges from 0 to 100, with higher score indicating worse symptom. The QLQ LC-13 is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30.
Pain score within 3 days after surgery (sub-study) | Up to 3 days after surgery
  Pain score is assessed with the Numeric Rating Scale, an 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality score within 3 days after surgery (sub-study) | Up to 3 days after surgery
  Subjective sleep quality is assessed with the Numeric Rating Scale, an 11-point scale where 0=the best sleep and 10=the worst sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Sullivan R, Alatise OI, Anderson BO, Audisio R, Autier P, Aggarwal A, Balch C, Brennan MF, Dare A, D'Cruz A, Eggermont AM, Fleming K, Gueye SM, Hagander L, Herrera CA, Holmer H, Ilbawi AM, Jarnheimer A, Ji JF, Kingham TP, Liberman J, Leather AJ, Meara JG, Mukhopadhyay S, Murthy SS, Omar S, Parham GP, Pramesh CS, Riviello R, Rodin D, Santini L, Shrikhande SV, Shrime M, Thomas R, Tsunoda AT, van de Velde C, Veronesi U, Vijaykumar DK, Watters D, Wang S, Wu YL, Zeiton M, Purushotham A. Global cancer surgery: delivering safe, affordable, and timely cancer surgery. Lancet Oncol. 2015 Sep;16(11):1193-224. doi: 10.1016/S1470-2045(15)00223-5. PMID 26427363
- [Background] Vansteenkiste J, Crino L, Dooms C, Douillard JY, Faivre-Finn C, Lim E, Rocco G, Senan S, Van Schil P, Veronesi G, Stahel R, Peters S, Felip E; Panel Members. 2nd ESMO Consensus Conference on Lung Cancer: early-stage non-small-cell lung cancer consensus on diagnosis, treatment and follow-up. Ann Oncol. 2014 Aug;25(8):1462-74. doi: 10.1093/annonc/mdu089. Epub 2014 Feb 20. PMID 24562446
- [Background] Emmert A, Straube C, Buentzel J, Roever C. Robotic versus thoracoscopic lung resection: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Sep;96(35):e7633. doi: 10.1097/MD.0000000000007633. PMID 28858083
- [Background] Ciechanowicz SJ, Ma D. Anaesthesia for oncological surgery - can it really influence cancer recurrence? Anaesthesia. 2016 Feb;71(2):127-31. doi: 10.1111/anae.13342. Epub 2015 Dec 16. No abstract available. PMID 26669960
- [Background] Kim R. Anesthetic technique and cancer recurrence in oncologic surgery: unraveling the puzzle. Cancer Metastasis Rev. 2017 Mar;36(1):159-177. doi: 10.1007/s10555-016-9647-8. PMID 27866303
- [Background] Byrne K, Levins KJ, Buggy DJ. Can anesthetic-analgesic technique during primary cancer surgery affect recurrence or metastasis? Can J Anaesth. 2016 Feb;63(2):184-92. doi: 10.1007/s12630-015-0523-8. PMID 26497721
- [Background] Mascha EJ, Yang D, Weiss S, Sessler DI. Intraoperative Mean Arterial Pressure Variability and 30-day Mortality in Patients Having Noncardiac Surgery. Anesthesiology. 2015 Jul;123(1):79-91. doi: 10.1097/ALN.0000000000000686. PMID 25929547
- [Background] Lonjaret L, Lairez O, Minville V, Geeraerts T. Optimal perioperative management of arterial blood pressure. Integr Blood Press Control. 2014 Sep 12;7:49-59. doi: 10.2147/IBPC.S45292. eCollection 2014. PMID 25278775
- [Background] Charlson ME, MacKenzie CR, Gold JP, Ales KL, Topkins M, Shires GT. Preoperative characteristics predicting intraoperative hypotension and hypertension among hypertensives and diabetics undergoing noncardiac surgery. Ann Surg. 1990 Jul;212(1):66-81. doi: 10.1097/00000658-199007000-00010. PMID 2363606
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Scholz AF, Oldroyd C, McCarthy K, Quinn TJ, Hewitt J. Systematic review and meta-analysis of risk factors for postoperative delirium among older patients undergoing gastrointestinal surgery. Br J Surg. 2016 Jan;103(2):e21-8. doi: 10.1002/bjs.10062. Epub 2015 Dec 16. PMID 26676760
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Younes RN, Rogatko A, Brennan MF. The influence of intraoperative hypotension and perioperative blood transfusion on disease-free survival in patients with complete resection of colorectal liver metastases. Ann Surg. 1991 Aug;214(2):107-13. doi: 10.1097/00000658-199108000-00003. PMID 1867517
- [Background] Park SY, Lee JG, Kim J, Bae MK, Lee CY, Kim DJ, Chung KY. The influence of smoking intensity on the clinicopathologic features and survival of patients with surgically treated non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):480-486. doi: 10.1016/j.lungcan.2013.07.002. Epub 2013 Jul 26. PMID 23896023
- [Background] Yu HC, Luo YX, Peng H, Wang XL, Yang ZH, Huang MJ, Kang L, Wang L, Wang JP. Association of perioperative blood pressure with long-term survival in rectal cancer patients. Chin J Cancer. 2016 Apr 11;35:38. doi: 10.1186/s40880-016-0100-8. PMID 27067550
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Bain CR, Draxler DF, Taylor R, Wallace S, Gouldthorpe O, Corcoran TB, Myles PS, L Medcalf R, Bozaoglu K. The early in-vivo effects of a single anti-emetic dose of dexamethasone on innate immune cell gene expression and activation in healthy volunteers. Anaesthesia. 2018 Aug;73(8):955-966. doi: 10.1111/anae.14306. Epub 2018 May 28. PMID 29806695
- [Background] Polderman JAW, Farhang-Razi V, van Dieren S, Kranke P, DeVries JH, Hollmann MW, Preckel B, Hermanides J. Adverse side-effects of dexamethasone in surgical patients - an abridged Cochrane systematic review. Anaesthesia. 2019 Jul;74(7):929-939. doi: 10.1111/anae.14610. Epub 2019 Mar 1. PMID 30821852
- [Background] Toner AJ, Ganeshanathan V, Chan MT, Ho KM, Corcoran TB. Safety of Perioperative Glucocorticoids in Elective Noncardiac Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2017 Feb;126(2):234-248. doi: 10.1097/ALN.0000000000001466. PMID 27922839
- [Background] Asehnoune K, Futier E, Feuillet F, Roquilly A; PACMAN group. PACMAN trial protocol, Perioperative Administration of Corticotherapy on Morbidity and mortality After Non-cardiac major surgery: a randomised, multicentre, double-blind, superiority study. BMJ Open. 2019 Mar 23;9(3):e021262. doi: 10.1136/bmjopen-2017-021262. PMID 30904834
- [Background] Call TR, Pace NL, Thorup DB, Maxfield D, Chortkoff B, Christensen J, Mulvihill SJ. Factors associated with improved survival after resection of pancreatic adenocarcinoma: a multivariable model. Anesthesiology. 2015 Feb;122(2):317-24. doi: 10.1097/ALN.0000000000000489. PMID 25305092
- [Background] Huang WW, Zhu WZ, Mu DL, Ji XQ, Nie XL, Li XY, Wang DX, Ma D. Perioperative Management May Improve Long-term Survival in Patients After Lung Cancer Surgery: A Retrospective Cohort Study. Anesth Analg. 2018 May;126(5):1666-1674. doi: 10.1213/ANE.0000000000002886. PMID 29517574
- [Background] Xu H, Shu SH, Wang D, Chai XQ, Xie YH, Zhou WD. Goal-directed fluid restriction using stroke volume variation and cardiac index during one-lung ventilation: a randomized controlled trial. J Thorac Dis. 2017 Sep;9(9):2992-3004. doi: 10.21037/jtd.2017.08.98. PMID 29221272
- [Background] Dinic VD, Stojanovic MD, Markovic D, Cvetanovic V, Vukovic AZ, Jankovic RJ. Enhanced Recovery in Thoracic Surgery: A Review. Front Med (Lausanne). 2018 Feb 5;5:14. doi: 10.3389/fmed.2018.00014. eCollection 2018. PMID 29459895
- [Background] Khwannimit B, Bhurayanontachai R. Prediction of fluid responsiveness in septic shock patients: comparing stroke volume variation by FloTrac/Vigileo and automated pulse pressure variation. Eur J Anaesthesiol. 2012 Feb;29(2):64-9. doi: 10.1097/EJA.0b013e32834b7d82. PMID 21946822
- [Background] Piccioni F, Bernasconi F, Tramontano GTA, Langer M. A systematic review of pulse pressure variation and stroke volume variation to predict fluid responsiveness during cardiac and thoracic surgery. J Clin Monit Comput. 2017 Aug;31(4):677-684. doi: 10.1007/s10877-016-9898-5. Epub 2016 Jun 15. PMID 27306799
- [Background] Suehiro K, Okutani R. Stroke volume variation as a predictor of fluid responsiveness in patients undergoing one-lung ventilation. J Cardiothorac Vasc Anesth. 2010 Oct;24(5):772-5. doi: 10.1053/j.jvca.2010.03.014. Epub 2010 Jul 17. PMID 20638869
- [Background] Zhang J, Chen CQ, Lei XZ, Feng ZY, Zhu SM. Goal-directed fluid optimization based on stroke volume variation and cardiac index during one-lung ventilation in patients undergoing thoracoscopy lobectomy operations: a pilot study. Clinics (Sao Paulo). 2013 Jul;68(7):1065-70. doi: 10.6061/clinics/2013(07)27. PMID 23917675
- [Background] Loop T. Fast track in thoracic surgery and anaesthesia: update of concepts. Curr Opin Anaesthesiol. 2016 Feb;29(1):20-5. doi: 10.1097/ACO.0000000000000282. PMID 26658180
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Detterbeck FC, Boffa DJ, Kim AW, Tanoue LT. The Eighth Edition Lung Cancer Stage Classification. Chest. 2017 Jan;151(1):193-203. doi: 10.1016/j.chest.2016.10.010. Epub 2016 Oct 22. PMID 27780786
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211